CLINICAL TRIAL: NCT05183737
Title: Effects of Supplementation With Microcapsules of Tumeric and Propolis on Inflammatory Markers in Patients on Hemodialysis
Brief Title: Effects of Microencapsulated Propolis and Turmeric in Patients With Chronic Kidney Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: DeniseMafra13
Record Dates: First submitted 2021-08-11; First posted 2022-01-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases; Inflammation
Keywords: Chronic Kidney Disease; Hemodialysis; Microcapsules; Inflammation; Propolis; Turmeric
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — Capsules; Curcumin; Propolis

STUDY DESIGN:
Intervention Model Description: The study is a longitudinal randomized, double-blind, placebo-controlled clinical trial with patients with CKD undergoing hemodialysis. Patients will be randomized and divided into two groups: intervention group, which will receive microcapsules containing 250mg of propolis and 250mg of turmeric, twice a day, for 12 weeks, and placebo group, which will receive for the same amount of capsules containing arabic gum and cornstarch.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microcapsules with turmeric and propolis (Active Comparator): Participants will receive microcapsules containing 0.250 milligrams of turmeric 95% curcumin and 0.250 milligrams of green propolis
  Interventions: Dietary Supplement: Microcapsules with turmeric and propolis
- Placebo Group (Placebo Comparator): Participants will receive microcapsules containing arabic gum and cornstarch with the same weight and characteristics as the intersecting microcapsules
  Interventions: Dietary Supplement: Microcapsules with turmeric and propolis

INTERVENTIONS:
Dietary Supplement: Microcapsules with turmeric and propolis — Participants will receive microcapsules containing 0.250 milligrams of turmeric 95% curcumin and 0.250 milligrams of green propolis, twice a day for 12 weeks

SUMMARY:
Oxidative stress and inflammation are correlated with Chronic Kidney Disease (CKD), in a way that they bring several harms to patients, including an increased risk of cardiovascular disease and mortality. Adjuvant therapeutic options such as bioactive compounds present in some foods seem to mitigate inflammation. Turmeric and propolis are foods that have compounds with antioxidant and anti-inflammatory capacity, as they promote the activation of nuclear erythroid transcription factor 2 (Nrf2 - responsible for the synthesis of antioxidant enzymes) and inhibit the activity of nuclear factor Kappa B (NF-κB - which increases the synthesis of inflammatory cytokines). This work aims to evaluate the effects of supplementation of associated propolis and turmeric microcapsules on inflammatory markers in patients with CKD undergoing hemodialysis (HD).

DETAILED DESCRIPTION:
The so-called Chronic Non-Communicable Diseases (NCDs) have been increasing in incidence. Among these, one can mention Chronic Kidney Disease (CKD). CKD is considered a public health problem and is characterized by an irreversible syndrome resulting from changes in the function or structure of the kidney, which has a progressive evolution.

Oxidative stress is one of the most potent inducers of inflammation, being an imbalance between the production of reactive oxygen species (ROS) and cellular antioxidant capacity, so that such imbalance can influence the activation of the nuclear factor kB (NF-κB), inflammation-associated interleukins, and tumor necrosis factor alpha 4 (TNF-α), which are promoters of cell damage and organic molecules. Patients with CKD on HD showed increased expression of NF-κB and reduced expression of Nrf2, so it is important to perform studies that propose ways to increase the performance of Nrf2, as well as reduce the activation of NF-κB. the performance of propolis and turmeric.

The study aims to evaluate the effects of supplementation of propolis and turmeric microcapsules on inflammatory markers and clinical parameters in patients with chronic kidney disease undergoing hemodialysis.

Sample calculation was performed using the G-Power 3.1 software, with a test power of 80%, considering the expression of NF-κB as the main outcome, significance level of 5% (two-tailed), effect size of 1, 32. The sample obtained consisted of 34 patients (17 in each group).

The proposed clinical study is a longitudinal randomized and double-blind (randomized controlled trial - RCT) where patients will receive capsules containing microencapsulated turmeric and propolis, twice a day, for 12 weeks. The mixture of microcapsules of propolis and turmeric will be distributed to participants in the form of hard gelatine capsules. The placebo group will receive the same amount of capsules, at the same times, containing gum arabic and corn starch. Randomization will be computerized in a 1:1 ratio.

* Anthropometric assessments, food intake, blood collections will be performed at the beginning of the follow-up and in subsequent consultations;
* The analysis of possible adverse effects will be collected through a separate analysis form;
* The assessment of food intake will be performed through the 3-day 24-hour recall;
* The assessment of nutritional status will be performed using anthropometric data;
* Blood samples will be collected in the morning, after fasting for 12 hours, before the dialysis procedure;
* NF-κB expression will be analyzed by means of peripheral blood nuclear cells (PBMCs) using real-time quantitative polymerase chain reaction (qPCR);
* For the measurement of inflammatory cytokines IL-6 and TNF-α, commercial ELISA kits will be used;
* C-reactive protein (CRP) will be determined by chemiluminescence;
* Lipid peroxidation will be estimated by determining thiobarbituric acid reactive substances (TBARS), including MDA, using the modified Ohkawa method;
* The evaluation of the total antioxidant capacity of the plasma will be determined by ELISA;

The effect of supplementation (∆) on each variable will be defined as the subject of the difference between the variable at the end of supplementation with propolis and turmeric and the value of the variable at the end of placebo administration. Statistical analyzes will be performed using SPSS version 22.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 5 CKD (GFR < 15 mL/min);
* On hemodialysis for more than 6 months;
* Who have arteriovenous fistula (AVF) as vascular access

Exclusion Criteria:

* Pregnant women;
* Smokers;
* Using antibiotics in the last 3 months;
* Using antioxidant supplements;
* Who have habitual intake of propolis, curcumin and turmeric;
* With autoimmune and infectious diseases, cancer, liver and AIDS (Acquired Immunodeficiency Syndrome)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The effects of the supplementation on the expression of transcription factors | 4 months
  Obtain blood samples to assess the effects of supplementation on biomarkers related to inflammation and antioxidant capacity, such as: erythroid nuclear transcription factor 2 (Nrf2) and nuclear factor Kappa B (NF-κB)
The effects of the supplementation on inflammatory cytokines | 4 months
  Get blood samples to evaluate the supplementation effects on cytokines (IL-6, TNF-α)

SECONDARY OUTCOMES:
The effects of supplementation on CRP levels | 4 months
  Measure before and after supplementation the levels of C-Reactive Protein (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mafra, phd, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No